CLINICAL TRIAL: NCT07156786
Title: N-Acetylcysteine Role on Urinary KIM-1 and Serum Creatinine Level in Cancer Patient With Cisplatin Based Chemotherapy
Brief Title: N-Acetylcysteine Roles in Preserving Renal Function Measured by Urinary KIM-1 (Kidney Injury Molecule-1) and Serum Creatinine on Cancer Patients With Cisplatin Based Chemotherapy: A Randomized Placebo-Controlled Trial
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, Oryza Gryagus Prabu, MD, Medical Staff, Internist, Fakultas Kedokteran Universitas Indonesia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-02-0179
Record Dates: First submitted 2025-08-24; First posted 2025-09-05 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Kidney Function Issue; Acute Kidney Injury; Cancer (Solid Tumors); Kidney Function Tests; Acetylcysteine Adverse Reaction
Keywords: kidney injury molecule 1; KIM-1; Creatinine; N-Acetylcysteine
MeSH Terms: conditions — Acute Kidney Injury; Neoplasms | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Patient receiving placebo and cisplatin chemotherapy
  Interventions: Drug: Placebo
- N-Acetylcysteine (Experimental): Patient receiving NAC + cisplatin based chemotherapy
  Interventions: Drug: N-acetylcysteine (NAC)

INTERVENTIONS:
Drug: N-acetylcysteine (NAC) — N-Acetylcysteine effercescent 1200 mg orally twice a day for 7 days. One day before cisplatin based chemotherapy, on the chemotherapy day, and five days after.
  Arms: N-Acetylcysteine
Drug: Placebo — Patient will get placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if N-Acetylcysteine drug works to protect kidney function in adults patient with cancer. Kidney function will be measured by laboratory parameter using urine sample (KIM-1 urine) and blood sample (serum creatinine). The main questions it aims to answer are:

1. Does N-Acetylcysteine lower the level of KIM-1 (Kidney Injury Molecule) in patients urine indicating kidney function protection?
2. Does N-Acetylcysteine lower the level of creatinine in patients blood indicating kidney function protection?

Participants will:

1. Had their blood and urine sample taken before taking the drugs (N-Acetylcysteine or placebo)
2. Underwent cisplatin based chemotherapy
3. Taken placebo or N-Acetylcysteine for seven days (1 day before chemotherapy, on the chemotherapy day, and 5 days after chemotherapy)
4. Had their blood and urine sample taken twice after taking the drugs (1 week and 3 weeks after chemotherapy)
5. Had their symptoms monitor during and after taking the drugs. Every possible side effect, hospitalization, or death will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cancer/ malignancy proven by histopathological examination
* Patient with GFR ≥60 ml/mins/1,73 m²
* Patient with normal complete blood count and liver function test result
* Patient with good performance status (Karnofsky score ≥80)
* Patients with cisplatin based chemotherapy

Exclusion Criteria:

* Patient that can not tolerate N-Acetylcysteine usage
* Patient with history of hypersensitivity to N-Acetylcysteine
* Patient that given other potentially nephrotoxic drug, such as furosemide, non-steroidal anti-infammatory drugs, aminoglycosides, amphotericin B, cephalosporine
* Patient that given other chemotherapy drug, such as permetrexed, ifosfamide, gemcitabin, bevacizumab, cetuxsimab
* Patient with history of malignant or uncontrolled hypertension
* patient with congestive heart failure, kidney structure abnormality, and acute infection
* Pregnant or lactating women
* Patient refusing to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Kidney injury molecule-1 | 1 week and 3 weeks after intervention
  Detected from participants urine sample indicating kidney function, will be measured at baseline, and after the intervention
Creatinine | 1 week and 3 weeks after intervention
  Creatinine will be measured from participants blood serum sample at baseline, and after intervention

IPD SHARING:
Plan to Share IPD: No
Due to privacy regulations and institutional policy, individual participant data will not be shared.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT07156786/Prot_SAP_000.pdf
  • Informed Consent Form (2025-09-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT07156786/ICF_001.pdf